CLINICAL TRIAL: NCT06668441
Title: A Phase I Pilot Clinical Trial of TNK Tissue-type Plasminogen Activator (rhTNK-tPA) Dose Escalation for Hypertension-Induced Intracerebral Hemorrhage Using Stereotactic Aspiration Technique to Remove the Hematoma
Brief Title: Minimally Invasive Surgery and RhTNK-tPA for Intracerebral Hemorrhage Evacuation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, deputy director, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-210
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Hemorrhages; Cerebrovascular Disorders; Cerebral Hemorrhage; Hemorrhage
Keywords: Basal ganglia; Stereotactic puncture therapy; Cerebral Hemorrhage; rhTNK-tPA; Minimally Invasive Surgery
MeSH Terms: conditions — Intracranial Hemorrhages; Cerebrovascular Disorders; Cerebral Hemorrhage; Hemorrhage | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teneplase assisted dissolution of blood clot therapy (Experimental): After CT reexamination 6 hours after surgery, the calculated injection amount of teneplase (teneplase injection amount = volume of hematoma × concentration of ascending drug) was diluted to 1ml with sterile injection water, and injected into the stereotaxically planned puncture path according to the location and size of the hematoma in turn. 0.5ml normal saline was used to flush the pipeline, and the drainage tube was fixed and closed for 2 hours. After the medication has fully acted with the hematoma mass, the drainage tube is re-opened to allow gravity drainage. CT examination was performed at 24 hours, 48 hours, 72 hours and 96 hours. Continuation or termination of the trial based on CT results at 24 hours, 48 hours, 72 hours, 96 hours: Teneplase was discontinued when the surgical goal defined by the test was achieved (residual hematoma ≤10ml), or new blood events occurred (compared with the previous time point CT, a CT value of > 72Hu and a volume of > 6ml of the space found in an
  Interventions: Drug: Minimally invasive surgery plus low-dose rhTNK-tPA group; Drug: Minimally invasive surgery plus medium dose rhTNK-tPA group; Drug: Minimally invasive surgery plus high dose rhTNK-tPA group

INTERVENTIONS:
Drug: Minimally invasive surgery plus low-dose rhTNK-tPA group — The calculated injection amount of teneplase (teneplase injection amount = volume of hematoma ×0.001mg) was diluted to 1ml with sterile injection water, and injected into the stereotaxically planned puncture path according to the location and size of the hematoma. The pipeline was rinsed with 0.5ml normal saline, and the drainage tube was fixed and closed for 2 hours, so that after the full effect of the drug on the hematoma mass was ensured. Re-open the drain to allow gravity drainage.
Drug: Minimally invasive surgery plus medium dose rhTNK-tPA group — The calculated injection amount of teneplase (teneplase injection amount = volume of hematoma ×0.003mg) was diluted to 1ml with sterile injection water, and injected into the stereotaxically planned puncture path according to the location and size of the hematoma. The pipeline was rinsed with 0.5ml normal saline, and the drainage tube was fixed and closed for 2 hours, so that after the full effect of the drug on the hematoma mass was ensured. Re-open the drain to allow gravity drainage.
Drug: Minimally invasive surgery plus high dose rhTNK-tPA group — The calculated injection amount of teneplase (teneplase injection amount = volume of hematoma ×0.009mg) was diluted to 1ml with sterile injection water, and injected into the stereotaxically planned puncture path according to the location and size of the hematoma. The pipeline was rinsed with 0.5ml normal saline, and the drainage tube was fixed and closed for 2 hours, so that after the full effect of the drug on the hematoma mass was ensured. Re-open the drain to allow gravity drainage.

SUMMARY:
The purpose of this trial is to determine the safety of using a combination of robot-assisted stereotactic puncture and clot lysis with rhTNK-tPA to remove intracerebral hemorrhage (ICH) and to provide dose evidence for a phase III clinical trial.

DETAILED DESCRIPTION:
Minimally invasive puncture surgery (MIPS) is a recommended effective surgical treatment method by the new guidelines to improve the mortality rate of intracerebral hemorrhage patients. It is easy to operate and has the conditions for widespread implementation. Stereotactic puncture is the least invasive treatment method, which can reduce the effect of hematoma occlusion and cytotoxicity and maximize the protection of neurological function. The MISTIE III study published in The Lancet showed that the mortality rate of the group treated with minimally invasive intracerebral hematoma evacuation combined with alteplase was reduced at 365 days, but the functional prognosis was not improved. Alteplase may have poor fibrin specificity, a short half-life, and a weak effect on PAI-1, resulting in incomplete blood clot dissolution, which may be the reason for poor prognosis. Tenecteplase (rhTNK-tPA), a third-generation specific fibrinolytic agent, is used for intravenous thrombolysis in acute ischemic stroke and has higher fibrin specifc. The study design is an open-label, non-comparative, phase 1 dose escalation protocol.The purpose of this trial is to determine the safety of using a combination of robot-assisted stereotactic puncture and clot lysis with rhTNK-tPA to remove intracerebral hemorrhage (ICH) and to provide dose evidence for a phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <80 years.
2. Symptoms must have manifested within 24 hours prior to the diagnostic CT scan. Cases with an indeterminate onset time are excluded. For patients who present symptoms upon sleeping, the last known time they were well should be used.
3. Acute spontaneous deep intracerebral hemorrhage (ICH) occurring in the basal ganglia or thalamus, with a volume between 20-50 mL as measured by ABC/2 method with radiographic imaging (CT, etc.).
4. Glasgow Coma Scale (GCS) score of 5-14.
5. Stability CT scan done at least 6 hours after diagnostic CT showing clot stability (growth <5 mL as measured by ABC/2 method).
6. Neuronavigation-assisted stereotactic MIPS should be performed within 6 to 24 hours after the diagnostic CT.
7. Systolic blood pressure (SBP) less than 180 mmHg maintained for a duration of six hours, documented proximate to the enrollment time point.

Historical Rankin score of 0 or 1.

Exclusion Criteria:

1. Lobar or subtentorial hemorrhage, including posterior fossa hemorrhage and cerebellar hemorrhage.
2. Stability CT scan done at least 6 hours after diagnostic CT showing clot instability (growth ≥5 mL as measured by ABC/2 method).
3. Intraventricular hemorrhage necessitating intervention to address mass effect or midline shift attributable to trapped ventricle syndrome secondary to intraventricular hemorrhage (IVH)-related casting.
4. Hemorrhage attributable to other cerebrovascular pathologies, including but not limited to ruptured aneurysm, arteriovenous malformation (AVM), vascular anomalies, moyamoya disease, hemorrhagic transformation of an ischemic infarct, or recurrence of a recent hemorrhage within the past year, as diagnosed through radiographic imaging.
5. Patients presenting with an unstable intracranial mass or progressive intracranial compartment syndrome.
6. Thalamic hemorrhages exhibiting evident extension into the midbrain, accompanied by oculomotor nerve palsy or pupils that are dilated and non-reactive. Other supranuclear gaze abnormalities do not constitute exclusion criteria.
7. Irreversible impairment of brainstem function, characterized by bilateral fixed and dilated pupils, extensor motor posturing, and a Glasgow Coma Scale (GCS) score of ≤ 4.
8. Indications for craniotomy in patients include: 1) progressive impairment of consciousness; 2) presence of brain herniation, with signs related to cerebellar tonsil herniation or temporal lobe gyrus herniation; 3) hematoma located within 1 cm of the cortical surface.
9. CT evidence suggesting a high risk of rebleeding, such as spot sign.
10. Platelet count <100,000/mL; INR >1.4.
11. Any irreversible coagulation disorders (e.g., hemophilia, von Willebrand disease, use of anticoagulants such as warfarin) or known clotting disorders (e.g., hypercoagulable states).
12. Inability to maintain INR ≤1.4 using short-acting and long-acting procoagulants (e.g., recombinant human coagulation factor VIIa, fresh frozen plasma, vitamin K, etc.).
13. Subjects necessitating long-term anticoagulation therapy are excluded from participation. Reversal of anticoagulation is permissible for medically stable patients who can feasibly tolerate the short-term risks associated with reversal. Patients must not require Coumadin (warfarin) or other anticoagulants during the initial 30-day period.
14. Prior to the onset of symptoms, anticoagulants such as dabigatran, apixaban, or rivaroxaban, as well as treatments like tirofiban, ticagrelor, cilostazol, or clopidogrel, were used.
15. Internal bleeding involving the retroperitoneal, gastrointestinal, or genitourinary system, or respiratory tract bleeding.
16. Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures, etc.) or site of recent surgical intervention.
17. Positive urine or serum pregnancy test in pre-menopausal female subjects without a documented history of surgical sterilization.
18. Allergy/sensitivity to TNK.
19. Engagement in a concurrent interventional clinical investigation or trial. Patients enrolled in observational, natural history, or epidemiological studies that do not involve any form of intervention remain eligible.
20. The presence of any concurrent serious illness that could confound outcome assessments, including but not limited to hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, or hematologic disorders.
21. Patients with mechanical heart valves are excluded. The presence of bioprosthetic valve(s) is permissible.
22. Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. Atrial fibrillation without mitral stenosis is permitted.
23. Any other condition that, in the investigator's judgment, would present a significant risk to the subject if the investigational therapy were to be initiated.
24. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
25. Patients deemed by the investigator to have unstable conditions that may benefit from other treatments.
26. Patients requesting conservative treatment or standard craniotomy microsurgery treatment.

The subject or their legal guardian/representative demonstrates an inability or lack of willingness to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Drug-related rebleeding events: | Within 24 hours of the last dose
  CT examinations were performed at 24, 48, 72, and 96 hours after administration. Compared with the CT at the previous time point, a CT value of more than 72 HU and a volume of more than 5 ml found in and around the hematoma cavity were defined as newly emitted blood.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- : Beijing Tongren Hospital, Capital Medical University,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou X, Chen J, Li Q, Ren G, Yao G, Liu M, Dong Q, Guo J, Li L, Guo J, Xie P. Minimally invasive surgery for spontaneous supratentorial intracerebral hemorrhage: a meta-analysis of randomized controlled trials. Stroke. 2012 Nov;43(11):2923-30. doi: 10.1161/STROKEAHA.112.667535. Epub 2012 Sep 18. PMID 22989500
- [Background] Wang WZ, Jiang B, Liu HM, Li D, Lu CZ, Zhao YD, Sander JW. Minimally invasive craniopuncture therapy vs. conservative treatment for spontaneous intracerebral hemorrhage: results from a randomized clinical trial in China. Int J Stroke. 2009 Feb;4(1):11-6. doi: 10.1111/j.1747-4949.2009.00239.x. PMID 19236490
- [Background] Scaggiante J, Zhang X, Mocco J, Kellner CP. Minimally Invasive Surgery for Intracerebral Hemorrhage. Stroke. 2018 Nov;49(11):2612-2620. doi: 10.1161/STROKEAHA.118.020688. PMID 30355183
- [Background] Li M, Mu F, Su D, Han Q, Guo Z, Chen T. Different surgical interventions for patients with spontaneous supratentorial intracranial hemorrhage: A network meta-analysis. Clin Neurol Neurosurg. 2020 Jan;188:105617. doi: 10.1016/j.clineuro.2019.105617. Epub 2019 Nov 20. PMID 31775069
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Background] Guo G, Pan C, Guo W, Bai S, Nie H, Feng Y, Li G, Deng H, Ma Y, Zhu S, Tang Z. Efficacy and safety of four interventions for spontaneous supratentorial intracerebral hemorrhage: a network meta-analysis. J Neurointerv Surg. 2020 Jun;12(6):598-604. doi: 10.1136/neurintsurg-2019-015362. Epub 2020 Jan 3. PMID 31900351
- [Derived] Wu Z, Wang M, Bai X, Tang J, Ni Y, Zhao S, Wang P, He Q, Huo R, Jiao Y, Wang D, Cao Y. Phase I dose-escalation study of tenecteplase, a third-generation fibrinolytic agent, combined with neuronavigation-assisted stereotactic minimally invasive puncture, in patients with acute spontaneous deep cerebral haemorrhage. Stroke Vasc Neurol. 2025 Sep 24:svn-2025-004389. doi: 10.1136/svn-2025-004389. Online ahead of print. PMID 40992931